CLINICAL TRIAL: NCT04657276
Title: Turkish Adaptation, Validity and Reliability of Segmental Assessment of Trunk Control (SATCo) Into in Infants With Down Syndrome
Brief Title: Turkish Adaptation of Segmental Assessment of Trunk Control Scale
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Esra Kınacı Biber, Research Assistant, Hacettepe University
Other Study IDs: GO 20/11
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2023-03

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Down Syndome: Infants with Down Syndrome

SUMMARY:
In infants with Down syndrome at risk in terms of neurosensory motor development retardation, the level of trunk control can determine the level of trunk control towards motor development in infants with down syndrome.

For this reason, the purpose of this study is to adapt the segmental assessment of trunk control scale to Turkish by evaluating the motor development in children with Down syndrome. It is the investigation of validity and reliability.

DETAILED DESCRIPTION:
Independent sitting of babies with Down syndrome is very important because sitting is the primary position on improving play activities. It is a known fact that late acquisition of sitting posture has negative effects on gross motor skills such as crawling and walking as well as fine motor skills. The extent to which trunk development affects the developmental stages of the child and his performance in motor behaviors and skills should be evaluated. At the same time, trunk control should be evaluated at various periods in order to determine early intervention and treatment strategies in babies with Down syndrome who are at risk for motor development.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer parents who have;
* Infant with down syndrome

Exclusion Criteria:

* Have a serious medical history (serious cardiac problems, infantile spasm, leukemia)
* Presence of MSS and PSS-related problems
* Those with visual and auditory problems
* Having epileptic seizures
* Presence of musculoskeletal problems

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Down Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Segmental Assesment of Trunk Control | 20 minutes
  It is an evaluation method that allows to evaluate the body control as static, active and reactive control, according to the body control levels. Examines the development of trunk control from level 1 (head control) and level 7 (full trunk control).
Gross Motor Function Measure (GMFM-88) | 30 minutes
  The Gross Motor Function Measure (GMFM) is an assessment tool designed and evaluated to measure changes in gross motor function over time or with intervention in children with cerebral palsy. tem scoring is the same for the GMFM-88. There is a scoring system with each item scored as 0, 1, 2, 3, or "not tested". A scoring key of 0 - does not initiate, 1 - initiates, 2 - partially completes, and 3 - completed, is used. High total score represents good development.

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory-PedsQL | 15 minutes
  PedsQL ™ Infant Scale
  On the PedsQL Generic Core Scales, for ease of interpretability, items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better HRQOL
Alberta Infant Motor Scale | 20 minutes
  Alberta Infant Motor Scale The total raw score is the sum of the scores for the four positions, which can range between 0 to 58; higher scores indicate better motor development. The total raw score is converted to an age-based percentile rank, varying from 5 to 90% for comparison norms

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Kınacı Biber, Ankara, Turkey (Türkiye)